CLINICAL TRIAL: NCT00766259
Title: Relationship of Staphylococcal Colonization to Infection
Status: Withdrawn | Type: Observational
Why Stopped: poor accrual
Sponsor: Veterans BioMedical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Eng-MRSA
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2021-03

CONDITIONS: MRSA Infection
Keywords: methicillin-resistant Staphylococcus; colonization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — only bacterial strains collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Hemodialysis
- 2: Intensive care
- 3: vascular patients with open wounds
- 4: nursing home
- 5: skin infections
- 6: control- ambulatory care clinic patients with no infections

SUMMARY:
Inpatients will be prospectively have nares screened and MRSA strains collected. All clinical MRSA strains of patients will also be prospectively collected. A sensitive strain discrimination test of spa typing will be used to determine if the strains are related. Hypotheses are

1. Strain colonization durations vary and may be very short in days to weeks.
2. Colonizing strains rarely infect 3) Both 1 and 2 may be affected by the patient's co-morbidity.

DETAILED DESCRIPTION:
Patients of special interest:

1. Skin and soft tissue infection
2. Nursing home patients
3. Vascular patients with leg lesions
4. ICU patients
5. Hemodialysis patients
6. Outpatients without history of infections(controls) will have nares screened for MRSA and then monthly for 1 year.

All strains will be saved and spa typed. Analysis of the data will be performed to answer the questions and hypotheses and to answer is the screening effort and the isolation of patients for MRSA as is in current practice worthwhile and is there any scientific data to support this practice

ELIGIBILITY:
Inclusion Criteria:

* Admitted and one of the co-morbid groups
* Ambulatory care patient with no infections

Exclusion Criteria:

* All others

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients admited
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Percent of infection strains which were also colonizer earlier | 3 years

SECONDARY OUTCOMES:
Duration of strain colonization among co-morbidity cohorts | 3 years